CLINICAL TRIAL: NCT02266290
Title: Effect of Kinesio® Taping on Measurements of Balance in Subjects With Chronic Ankle Instability: a Randomized Clinical Trial
Brief Title: Effect of Kinesio® Taping in Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URJC_21_2012
Record Dates: First submitted 2014-10-10; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Ankle Sprain
Keywords: ADHESIVE TAPE; ANKLE INJURY; POSTURAL BALANCE; FUNCTIONAL ANKLE INSTABILITY
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kinesio-Tape group (Experimental): In this study, Sport tex® kinesiotape over lateral ankle (6cm*2.5m) is used.
  Interventions: Procedure: taping of ankle sprain; Device: Sport tex® kinesiotape
- Placebo Tape Group (Placebo Comparator): In the placebo group, Pretape Cramer® (100% cotton, 1.25cm*10m) was used. With patient in the same position described above, horizontal strips were placed covering the sural region with no defined direction.
  Interventions: Procedure: taping of ankle sprain; Device: Pretape Cramer®

INTERVENTIONS:
Procedure: taping of ankle sprain — All participants were taped for a lateral ankle sprain. The individual is in supine position keeping the foot and ankle in a neutral position. The strip (I) is applied with not stretch in the outside of the leg just above the ankle, and then the rest of the strip is applied on the outside of the ankle and under the heel.
Device: Sport tex® kinesiotape
  Arms: Kinesio-Tape group
Device: Pretape Cramer®
  Arms: Placebo Tape Group

SUMMARY:
The Objective is to examine the immediate and prolonged effects (seven days) of Kinesio® Tape (KT) on balance in subjects with chronic ankle instability using Computerized dynamic posturography (CDP). Design. A 7 days follow-up, single-blind randomized controlled trial. Setting. University community. Participants. A sample of 30 subjects aged 18 to 28 with CAI and subjective perception of ankle instability (FAI) was enrolled in this study. Interventions. Participants will be randomly divided into two groups: an experimental group in which was applied KT, and a control group in which was applied a placebo tape.Objective. To examine the immediate and prolonged effects (seven days) of Kinesio® Tape (KT) on balance in subjects with chronic ankle instability using Computerized dynamic posturography (CDP). Design. A 7 days follow-up, single-blind randomized controlled trial. Setting. University community. Participants. A sample of 30 subjects aged 18 to 28 with CAI and subjective perception of ankle instability (FAI) was enrolled in this study. Interventions. Participants were randomly divided into two groups: an experimental group in which was applied KT, and a control group in which was applied a placebo tape. Main Outcome Measure(s). The CDP device employed in this study was Smart Equitest® version 8.2. CDP analysis was conducted using the Sensory organization test (SOT). The composite SOT score (COMP) and the composite SOT strategy (STR), the partial score for SOT condition 2 (SOT 2) and its strategy (STR 2) were considered as outcomes measures.

DETAILED DESCRIPTION:
Participants were randomly distributed (using the QuickCalcs application from GraphPad Software)a into two groups: an experimental group in which was applied KT, and a control group in which was applied a placebo tape. All outcomes in both groups were assessed by an assessor blinded to the subject´s allocation. Individuals were also blinded to the allocation group. Balance was assessed using the SOT under three conditions: (1) without taping; (2) immediately following application; (3) following 7 days of use.

Computerized dynamic posturography is used to measure the balance. Subjects had to maintain their COG stable in 3 consecutive series of 20s duration for each of the 6 conditions in the test. In the first 3 conditions, the platform remained fixed. Condition 1 was conducted with open eyes, condition 2 with closed eyes and condition 3 with a mobile visual environment referenced to postural oscillations. Conditions 4, 5 and 6 repeated the visual conditions of the first 3 tests and added platform movement referenced to the anteroposterior oscillation of the subject, with the ankle-foot angle remaining constant, thus annulling proprioceptive sensory input.

The system utilizes force-plate technology (two 23 × 46 cm footplates) to determine the location of the COG within predefined 75% limits of stability while adjusting for an individual subject's height (COG = 0.55 × height). For each test, the software provides measures of postural sway and the ability to maintain the COG within a predefined target area resulting in partial scores for each condition and an overall balance score (composite SOT score, COMP) (%). The theoretical maximum displacement a normal subject may sway without fall is assumed to be 12.5 degrees (8.25 degrees anterior, 4.25 degrees posterior). The equilibrium score = 12.5 - Ɵ (maximum - minimum)/12.5 × 100%, where Ɵ is the maximum anteroposterior COG sway angle recorded in each trial. Values close to 100% indicated minimum balancing. Test was scored with a value of 0 when patients needed help or took a step to maintain balance.

SOT condition 2 is the best trial in order to assess the influence of KT on proprioceptive system in subjects without vestibular deficits. As primaries outcome measures, the composite SOT score (COMP) and the composite SOT strategy (STR), were chosen. The partial score for SOT condition 2 (SOT 2) and its strategy (STR 2) were considered as secondary outcomes measures. SOT condition 2 is carried out with closed eyes. Therefore, balance under this condition is controlled mainly by the proprioceptive system, in which, according several authors, KT could have an effect. Under these All subjects were initially familiarized with the CDP before undergoing. Multiple baseline measures of the SOT were administrated in order to document change due to tape application and to avoid the learning effect.26 It has been suggested a short-term adaption that reduces the postural sway by either increasing the stiffness in the ankles or through reweighting of sensory information.

ELIGIBILITY:
Inclusion Criteria:

* history of at least 1 acute lateral ankle sprain that resulted in swelling, pain, and temporary loss of function (but none in the previous 3 months).
* history of multiple episodes of the ankle ''giving-way'' in the past 6 months-
* a score below 27 in the Cumberland Ankle Instability Tool.
* evidence of mechanical instability assessed by a physician using an anterior drawer test

Exclusion Criteria:

* history of lower limb injury other than the unilateral Chronic ankle instability and skin allergy to the tape.
* To be actively involved in any kind of physical activity or rehabilitation program.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Computerized dynamic posturography | 7 days
  The CDP device employed in this study was Smart Equitest® version 8.2 (NeuroCom International Inc., Clackamas, OR, USA). Posturography analysis was conducted using the SOT. This test assesses postural control through the use of external stimuli on the visual and proprioceptive system.
  Participants were instructed to stand on the force-plate facing the visual surround. A safety harness was fixed to prevent injury from falls. Their bare feet position on force-plates was adjusted according to the height of the patient, as marked on the equipment. Subjects had to maintain their COG stable in 3 consecutive series of 20s duration for each of the 6 conditions in the test.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Mª Alguacil-DIego, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Francisco Molina Rueda. Avda. de Atenas. s/n., Alcorcón, Madrid, Spain

REFERENCES:
- [Derived] de-la-Torre-Domingo C, Alguacil-Diego IM, Molina-Rueda F, Lopez-Roman A, Fernandez-Carnero J. Effect of Kinesiology Tape on Measurements of Balance in Subjects With Chronic Ankle Instability: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2015 Dec;96(12):2169-75. doi: 10.1016/j.apmr.2015.06.022. Epub 2015 Sep 7. PMID 26360974
- See also: University — http://www.urjc.es